CLINICAL TRIAL: NCT02925481
Title: Yoga Online: Interconception Care to Prevent PTSD Symptoms After Stillbirth
Brief Title: Yoga Online Feasibility to Reduce PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Huberty, Associate Professor in the School of Nutrition and Health Promotion, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34AT008808 (NIH); R34AT008808 (NIH)
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: PTSD
Keywords: Yoga; PTSD; mental health; stillbirth
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being; Stillbirth

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Low dose Yoga (Experimental): 12 week online yoga for 60 minutes per week
  Interventions: Behavioral: Low dose online yoga participation
- Moderate dose Yoga (Experimental): 12 week online yoga for 150 minutes per week
  Interventions: Behavioral: Moderate Online yoga participation
- Stretch and toning (Active Comparator): 12 week online stretching, toning exercises for 60 minutes per week
  Interventions: Behavioral: Stretching and toning

INTERVENTIONS:
Behavioral: Moderate Online yoga participation — Phase 1: Testing yoga videos for emotional regulation and self-compassion which will inform the selected videos for Phase 2 prescription Phase 2: 150 minutes of Online streaming yoga videos completed at home. Week 1/2 introductory videos that include short video clips breaking down each pose Weeks 3-12 increase in difficulty (all videos are appropriate for beginners)
  Other Names: MD
  Arms: Moderate dose Yoga
Behavioral: Stretching and toning — Phase 1: Developing 12 week prescription for online control videos Phase 2: Online streaming stretching and toning videos completed at home which consist of a warm-up, 1 balance, 2 core, 2-3 upper body and lower body exercises, 6 stretches, cool-down
  Other Names: STC
  Arms: Stretch and toning
Behavioral: Low dose online yoga participation — Phase 1: Testing yoga videos for emotional regulation and self-compassion which will inform the selected videos for Phase 2 prescription Phase 2: 60 minutes of Online streaming yoga videos completed at home. Week 1/2 introductory videos that include short video clips breaking down each pose Weeks 3-12 increase in difficulty (all videos are appropriate for beginners)
  Other Names: LD
  Arms: Low dose Yoga

SUMMARY:
Each year more than 26,000 pregnancies in the United States end in stillbirth (late fetal death at >20 weeks of gestation). A 2011 issue of the Lancet, dedicated entirely to stillbirth, recognized it as a "too-often-ignored" public health problem despite occurring once in every 160 pregnancies. The death of a baby is highly traumatic and can incite negative mental, emotional, and physical health consequences lasting years after the loss. Bereaved mothers with stillbirth have a 4-fold higher risk of depression and 6-fold higher risk for post-traumatic stress disorder (PTSD). These mental health consequences are likely to negatively affect subsequent pregnancies, many of which occur within the first year after loss (50-98%).

Inter-conception care is provided to women of reproductive age between pregnancies; however, few interventions focus on PTSD symptomatology and its related comorbidities in bereaved mothers. Treatment for bereaved mothers may include psychiatric medication and/or referral to support groups. Because bereaved mothers with stillbirth may have additional mental and physical health risks, pharmacological interventions are typically a first and sole line of treatment and may not sufficiently allay bereaved mothers' emotional distress. Moreover, women may be trying to conceive or may have already conceived and report reticence to taking medication. Additionally, support groups with little emphasis on coping may not be helpful for some grieving mothers.

Non-pharmacological approaches, such as yoga, may be an alternative option for bereaved women with stillbirth. Yoga has been established as an effective, safe, acceptable, and cost effective approach to improving mental health in a variety of populations, including pregnant and post-partum women. Yoga has also been used as a means to cope with PTSD associated with surviving a traumatic event (i.e., interpersonal violence, military veterans). The investigators are unaware of any studies that have explored yoga to reduce PTSD in bereaved mothers with stillbirth. Furthermore, online streaming yoga (on-demand videos played in the home) has recently grown in popularity and may address the unique barriers that women experiencing stillbirth may have. To reduce PTSD symptoms and its co-morbid conditions (i.e., anxiety and depression) the investigators propose to develop and test the feasibility and acceptability of a home-based, online streamed yoga intervention (www.udaya.com) for bereaved mothers with stillbirth.

DETAILED DESCRIPTION:
Phase 1 (pre-recruitment):

Racial/ethnic panel:

The investigators will recruit a panel of racial/ethnic minority women (African American and Hispanic women) who have experienced stillbirth (n=5) and discuss potential benefits and perceptions of yoga to inform the study. Women will be asked to complete a web-based eligibility and informed consent survey via Qualtrics. In addition, the investigators will inquire on ways to encourage enrollment of racial/ethnic minority women into the study. The investigators will use this information to potentially modify recruitment materials in phase 2. If modification for recruitment materials are needed based on interviews, the investigators will submit the modifications to the IRB at that time. Interviews will take approximately 15-20 minutes and will be conducted over the phone.

Iterative design process for yoga prescription: Before the investigators begin recruitment for the study the investigators will implement the following steps to determine the yoga prescription for the LD and MD intervention groups:

1. Identify videos from existing Udaya library. Videos prescribed will be selected for qualities pertaining to selected potential mechanisms proposed in our conceptual model. Classes chosen will include detailed instruction and specific alignment cues to promote focus and attention, thus potentially reducing sensitivity to internal sensations and increase affect tolerance (emotional regulation) (e.g., press your hands into the mat in cobra pose, lift your toes during chair pose). Also slow moving classes with longer holds to encourage non-reactivity and awareness of negative thoughts or self-criticism.
2. Gather a panel of women who have experienced stillbirth (n=5) and a panel of women who regularly do yoga (n=5) to review the videos (including, as appropriate, engaging in practices. Women will be asked to complete a web-based eligibility survey and informed consent via Qualtrics. Each woman will review ~9 yoga videos within a 6 week period (videos outlined in #1). Women will be asked to come into the Healthy Lifestyles Research Lab at Arizona State University on a weekly basis for 6 weeks (1-2x/week). Before and after the review, the team will actively explore if individuals feel they are connected to their body, feel emotionally regulated, and self-compassionate (see #3 below). Sessions not perceived as useful for self-compassion and emotional regulation will be replaced for the proposed study. If no previously developed videos are supportive of improving self-compassion and emotional regulation, the investigators will produce new classes (up to six 30-min classes) in partnership with Udaya.
3. Have participants rate their current self-compassion and emotional regulation to gather the pre-post mean score changes for all videos. This pre-post questionnaire will take roughly 5 minutes to complete. The investigators will also ask questions during post-intervention interviews to glean further insights about the utility of the yoga sessions for improving self-compassion and emotional regulation. This process will inform the videos to be used in the future larger trial Phase 2.

For our purposes, all classes for the intervention will be screened for applicability by the yoga therapist. Participants' username and passwords will provide them access to only the yoga videos prescribed; participants will not have access to the complete Udaya library of yoga videos. Participants will be asked to complete the yoga videos in a specific order, which will include specialized preparatory instructions for each class to quell apprehension and further ensure safety.

After this process the investigators will finalize the yoga prescription for Phase 2 and will submit any modifications to the IRB before recruitment begins.

Phase 2 Enrollment: Interested participants will complete an eligibility screener on a Qualtrics link, or contact the research team via phone or email. Our current screener takes approximately 5-10 mins to complete. Research team members will follow a script to respond to interested participants who phone or email, and refer them to the eligibility screener. Eligible participants will receive an email requesting times to schedule a 15 minute intake call (i.e., explain the study) and an email confirmation for the appointment. Following the intake appointment, eligible participants will receive a Qualtrics link asking them to electronically sign an informed consent and participate in a baseline assessment of self-report measures that will take approximately 20 minutes. After this step, participants will be randomized to intervention or control group (See below). Ineligible participants will be notified by phone and offered a discounted Udaya.com membership.

Randomization: The investigators will randomize participants into low dose intervention group (LD; n=30), moderate dose intervention group (MD; n=30), or stretch and tone control group (STC; n=30) after the informed consent and baseline questionnaires have been complete. Research personnel will use a computer-generated list of numbers (i.e., randomizer.org). Research personnel who assign participants to a group will not be the same as those who download or clean data. Additionally, group status will be entered separately so that research personnel downloading data will be blinded to treatment assignment. Women in LD and MD will be prescribed 60 mins or 150 mins of yoga per wk respectively, for 12 wks. The STC group will complete a minimum of 60 mins/wk of stretching/toning exercises to match LD intervention group.

Tracking. Participation in the videos for all groups (LD, MD, STC) will be tracked (class taken, time of day, length of use etc.) on the Udaya.com website throughout the study. Before beginning the study, the research team will send each participant a daily log Qualtrics link to self-track: (a) completion of yoga/stretching sessions; (b) rate of perceived exertion; (c) assessment of mindfulness; (d) other PA participation; (e) participation in psychotherapy (i.e., cognitive behavioral therapy); and (f) pregnancy, mental health, and use of psychiatric medication (see daily/weekly log). Research personnel will contact participants weekly (via email/text) to remind them to participate in yoga/stretching and complete daily/weekly logs. Participants will be given a choice of text or email reminders. If a participant from the intervention or STC is not meeting their minimal dose requirement and/or not tracking their sessions, research personnel will reach out to the participant via text/email reminder.

Control (STC). The investigators will inform the adaptation of the STC group using Consultant McAuley's well established, evidence-based control group originally designed for older adults. The investigators will modify the prescription for the control group to be more age and population specific for the proposed study. All videos will be produced by Udaya.com and taught by a trained exercise professional. The STC group will complete a minimum of 60 mins/wk of stretching/toning exercises to match the LD intervention group. The instructor will ask participants to perform each isolated stretch, limbering, or toning exercise for 20-30 seconds and repeat five times. Participants will be asked to perform slow, controlled, and complete movements. Women will be given 4 upper body, 4 lower body, 3 trunk/core, and 1-2 balance exercises, with appropriate progression over 12 wks. Retention of women in the control group is important to the internal validity of the study. As such, the stretch, limbering, and toning exercises will be combined in different orders within each video to prevent boredom as recommended by Consultant McAuley. An important adaptation for the control group is the provision of modifications of each individual exercise. For each exercise, the instructor will demonstrate a modified version that is slightly less difficult and a more challenging version that adds difficulty for those who have mastered the movement capabilities, these modifications will allow the program to be highly adaptable for women with a wide range of capabilities.

The STC videos will have discussion related to form and safety by the instructor (i.e., no guidance for movement with breath or mindfulness). Additionally, videos will have students in the background following instructor cues and demonstrating variations of exercises. There will be no final relaxation pose in the STC videos (i.e., the rest period during which the efforts of PA are soothed, the mind is most receptive to stillness, and the cultivation of mindfulness culminates). Usernames and passwords for women in the control group will be specific to accessing only the STC group videos on Udaya.com.

Pregnancy during Intervention:

In the case that a woman becomes pregnant during this study the investigators will ask her to complete the Physical Activity Readiness Medical Examination for Pregnancy (PARmed-X for Pregnancy), a health-screening tool for participation in prenatal exercise. The PARmed-X for pregnancy is completed with their primary care physician to identify any contraindications to exercise, and includes 29 questions pertaining to general health status, status of current pregnancy, physical activity habits over the last month, and absolute and relative contraindications.

It has been well established that yoga is safe during pregnancy and postpartum and all classes prescribed will be suitable for women up to 20-wks gestation (the maximum possible based on our study eligibility). At any time during the study, if the participant's medical team advise her not to participate in yoga or other exercise, she would be immediately withdrawn from the study. Pregnancy status will be tracked throughout the 12-week study period via weekly assessment in weekly logs.

Post-intervention:

Post-intervention questionnaires will be administered via web-based survey (i.e., Qualtrics) at the end of week 12. In addition, follow-up surveys will be administered via web-based survey (i.e., Qualtrics) at 20-wks post baseline assessments.

Qualitative interviews following best practices for conducting interviews will be conducted with 15 participants. The qualitative interviews will be used to supplement information gained from the satisfaction surveys and to further understand the use of non-pharmacological interventions such as yoga in this population. Purposive sampling strategies (i.e., maximum variation sampling) will be used to understand individuals' experiences and inform the future larger trial. The investigators will specifically select participants from the study (approximately 5 from each intervention group, and 5 from control group or until data saturation has been reached) that represent those who had high/low compliance (at least 3 of 5 will be those who had low compliance (i.e., not reaching their prescribed minimal dose of yoga) and at least 3 of 5 will be racial/ethnic minorities). Qualitative interviews will be administered in the intervention groups at post-intervention (12 wks) and at follow-up (20 wks) and will last approximately 15-20 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Women who experienced stillbirth (>20 wks gestation) within past 24 mos
2. Clinical levels posttraumatic stress symptoms (>33 as measured by the IES-R)
3. ≥ 18 yrs of age
4. Residing in U.S.
5. Able to read/understand English
6. Underactive (≤120 mins/wk moderate intensity PA)
7. Willing to be randomized
8. Answer "no" to all items on PA Readiness Questionnaire (can participate safely), or if a woman answers "yes" to one or more questions on the PAR-Q, she will be asked to obtain medical clearance from her physician prior to participation in the study. Women will be given two options in which to demonstrate medical clearance (a) bring a form provided by the study team to their health care provider to obtain a signature from a physician and then email, fax, or mail the signed medical clearance form to the research personnel, or (b) sign and fax a release of information form to research personnel, who will then send the medical clearance form directly to their designated health care providers' office to obtain a physician signature.

Exclusion Criteria:

1. Unstable psychiatric condition (psychosis; suicidal ideation with plan)
2. Pregnant at time of enrollment
3. Practicing yoga at least 60 mins/wk
4. Unwilling to be randomized to a group.
5. At risk for suicide based on follow-up phone assessment by a trained contact person under supervision of Dr. Cacciatore after positive screen
6. (PHQ-9 score of 1, 2, or 3)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Clinically elevated levels of PTSD (according to IES-R) | 12 weeks

SECONDARY OUTCOMES:
Impact of Events Survey (IES-R) | 12 weeks post baseline
  Post-traumatic stress disorder symptoms were measured using the Impact of Events Scale (IES-R). The IES-R was developed to reflect the criteria for PTSD per the Diagnostic Symptom Manual (DSM-IV). There scale consists of 22 questions which are scored on a five-point Likert scale (0=not at all, 1=a little bit, 2=moderately, 3=quite a bit, 4=extremely). There are three subscales (i.e., avoidance, intrusion, hyperarousal) and the sub of the three subscales scores comprise the total score. A total score ≥33 indicates the likely presence of PTSD.
State-Trait Anxiety Inventory | 12 weeks post baseline
  The State-Trait Anxiety Inventory (STAI) yields scores indicating levels of train (Form Y-1) and state (Form Y-2) anxiety, with higher scores indicating greater levels of anxiety. This scale is scored using a four-point Likert scale(1=not at all, 2=somewhat, 3=moderately so, 4=very much so), and participants respond to questions such as, "I feel calm," and "I feel nervous and restless." The STAI has demonstrated reliability in pregnant and postpartum populations.
Patient Health Questionnaire (PHQ-9) | 12 weeks post baseline
  The Patient Health Questionnaire-9 (PHQ-9) was used to measure depressive symptoms. This measure is commonly used to screen, diagnose, monitor, and measure the severity of depression, Scores range from 0-27 and cut-off scores of 5, 10, 15, and 20 indicate mild, moderate, moderately severe, and severe depressive symptoms, respectively. This scale is valid and reliable in general populations (α=.86-.89) and has been validated in pregnant and postpartum populations.
Perinatal Grief Scale (PGS) | 12 weeks post baseline
  The Perinatal Grief Scale (PGS) is a valid 33-item instrument used to quantify the grief of perinatal loss. This scale consists of three subscales (active grief, difficulty coping, and despair) and uses a 5-point Likert scale (1=strongly agree to 5=disagree). The three subscales have a possible range of 11-55, and higher scores indicate more intense grief.
Self-Compassion Scale | 12 weeks post baseline
  The Self-Compassion Scale (SCS) is a 26-item questionnaire using a five-point Likert scale from 1=almost never to 5=almost always, The SCS consists of six subscales (self-kindness, self-judgment, common humanity, isolation, mindfulness, over-identified) and has good construct validity and reliability (α=.92). A total score is calculated by taking the mean of each subscale and reverse scoring the negative subscale items (i.e., self-judgment, isolation, over-identification) and computing a total mean. Higher scores indicate higher levels of self-compassion. A sample question includes, "When times are really difficult, I tend to be tough on myself."
Emotional Regulation Questionnaire (ERQ) | 12 weeks post baseline
  The Emotion Regulation Questionnaire (ERQ) is a 10-item scale used to measure an individual's tendency to regulate his or her emotions by two strategies: cognitive reappraisal and expressive suppression. Higher scores indicate greater use of emotional regulation strategies.
Pittsburgh Sleep Quality Index | 12 weeks post baseline
  Sleep was measured subjectively using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-item questionnaire that has demonstrated reliability and validity in pregnant populations. Higher global PSQI scores indicate more sleep disturbances. We also measured sleep using objective measures.
Modifiable Activity Questionnaire (MAQ) | 12 weeks post baseline
  The Modifiable Activity Questionnaire (MAQ) is a self-report scale used to assess frequency and duration of various activities. It was designed to be modified to assess physical activity in different populations.
SF-12v2 Health Survey (SF-12) | 12 weeks post baseline
  The SF-12 is a 12-item scale assessing self-reported health. The scale was developed for and widely used in the general population. It is comprised of subscales with physical and mental health domains. The physical and mental composite sub-scores are scored on a scale from 0 (lowest level of health) to 100 (highest level of health).
Mindfulness Attention Awareness Scale (MAAS) | 12 weeks post baseline
  The Mindful Attention Awareness Scale (MAAS) is a 15-item scale that measures the extent to which individuals are able to maintain awareness of present-moment experience. This scale uses a 6-point Likert scale (ranging from 1=almost always to 6=almost never), and the mean is computed to generate a total score. Higher scores indicate higher levels of mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Huberty J, Sullivan M, Green J, Kurka J, Leiferman J, Gold K, Cacciatore J. Online yoga to reduce post traumatic stress in women who have experienced stillbirth: a randomized control feasibility trial. BMC Complement Med Ther. 2020 Jun 5;20(1):173. doi: 10.1186/s12906-020-02926-3. PMID 32503517
- [Derived] Huberty J, Matthews J, Leiferman J, Cacciatore J, Gold KJ. A study protocol of a three-group randomized feasibility trial of an online yoga intervention for mothers after stillbirth (The Mindful Health Study). Pilot Feasibility Stud. 2017 Jul 6;4:12. doi: 10.1186/s40814-017-0162-7. eCollection 2018. PMID 28694991